CLINICAL TRIAL: NCT01004796
Title: Estrogen-Related Receptor Alpha As A Novel Biomarker For Breast Cancer
Brief Title: Study of Biomarkers in Tissue Samples From Patients With Breast Cancer
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Other Study IDs: CDR0000357299; P30CA014520 (NIH); WCCC-CO-TEMP
Record Dates: First submitted 2009-10-29; First posted 2009-10-30 (Estimated); Last update posted 2016-02-29 (Estimated); Status verified 2016-02

CONDITIONS: Breast Cancer
Keywords: breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Cytogenetic Analysis; Microarray Analysis; Immunohistochemistry; Immunologic Techniques; Mass Spectrometry

INTERVENTIONS:
Genetic: cytogenetic analysis
Genetic: microarray analysis
Genetic: mutation analysis
Other: immunohistochemistry staining method
Other: immunologic technique
Other: mass spectrometry

SUMMARY:
RATIONALE: Studying samples of tumor tissue from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer.

PURPOSE: This research study is looking at tissue samples from patients with breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Identify by mass spectroscopy and site-specific mutagenesis the post-translational modifications of estrogen-related receptor alpha (ERRα1) that are responsible for ERRα1 function as a constitutive activator rather than a down-modulator of transcription of estrogen response element-regulated genes in tumors of patients with breast cancer.
* Produce a panel of monoclonal antibodies to ERRα1 by standard hybridoma methods that can be used to distinguish between the activator and repressor forms of this receptor in these patients.
* Validate the utility for immunohistochemistry (IHC) assays of some of the ERRα-specific sera by performing IHC and quantitative real-time PCR on some primary breast carcinomas.
* Correlate the results of IHC studies on archival paraffin sections of primary breast tumors using monoclonal antibodies to ERRα1, ERRα1 status, currently assayed biomarkers, and course of treatment with patient outcomes.

OUTLINE: Breast tumor tissue samples are obtained from a tissue bank in the form of frozen tumors and paraffin-embedded sections on microarray blocks. Monoclonal antibodies (MOABs) to ERRα1 are produced using antigens in these tissue samples and immunohistochemical studies are performed using the MOABs. Cytogenetic studies are performed on DNA purified from these tissue samples.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of breast cancer
* Tumor tissue available
* The following clinical information must be known:

  * ErbB2 status
  * Nodal status
  * Percent S phase
* Hormone receptor status:

  * Estrogen receptor and progesterone receptor status known

PATIENT CHARACTERISTICS:

* Menopausal status not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Max Age: 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult

PRIMARY OUTCOMES:
Post-translational modifications of estrogen-related receptor alpha (ERRα1) that are responsible for ERRα1 function as a constitutive activator rather than a down-modulator of transcription of estrogen response element-regulated genes
Production of a panel of monoclonal antibodies to ERRα1 by standard hybridoma methods that can be used to distinguish between the activator and repressor forms of this receptor
Validation of the utility for immunohistochemistry (IHC) assays of some of the ERRα-specific sera by performing IHC and quantitative real-time PCR on some primary breast carcinomas
Correlation of the results of IHC studies on archival paraffin sections of primary breast tumors using monoclonal antibodies to ERRα1, ERRα1 status, currently assayed biomarkers, and course of treatment with patient outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Janet E. Mertz, PhD, Study Chair — University of Wisconsin, Madison